CLINICAL TRIAL: NCT04813003
Title: How Altered Gut-Brain-Axis Influences Food Choices. (BrainFood) Part 1: Brain Imaging and Computational Modelling
Brief Title: How Altered Gut-Brain-Axis Influences Food Choices: Part 1
Acronym: BrainFood
Status: Completed | Type: Observational
Sponsor: Lia Bally (Other)
Collaborators: ETH Zurich (Other)
Responsible Party: Sponsor-Investigator, Lia Bally, Professor, Insel Gruppe AG, University Hospital Bern
Organization: Insel Gruppe AG, University Hospital Bern (Other)
Other Study IDs: BrainFood Part 1
Record Dates: First submitted 2021-01-18; First posted 2021-03-24 (Actual); Last update posted 2022-09-23 (Actual); Status verified 2022-09

CONDITIONS: Obesity; Food Preferences
Keywords: Obesity; Bariatric Surgery; Food Preferences; Food Behaviour; Computational Modelling; Functional Brain Imaging
MeSH Terms: conditions — Obesity; Food Preferences | interventions — Functional Neuroimaging

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Obesity group (group 1): Pilot phase:
  5 adults with class II-III obesity (BMI≥35kg/m2) planned for bariatric surgery will undergo functional imaging and neurobehavioural tasks before bariatric surgery.
  Refined protocol phase:
  20 overweight adults (BMI≥30kg/m2 or BMI≥28kg/m2 with adiposity-related comorbidities (prediabetes, type 2 diabetes mellitus, hypertension, dyslipidemia)), referred for obesity treatment (surgical or non-surgical).
  Interventions: Other: Functional Brain Imaging and neurobehavioural tasks
- Control group (group 2): Pilot phase:
  5 healthy adults with normal body mass (BMI 18.5-24.9kg/m2) matched for age-, sex- and education will serve as a control group and undergo the same experiment.
  Refined protocol:
  20 healthy adults with normal body mass (BMI 18.5-24.9kg/m2) matched for age and sex will serve as a control group and undergo the same experiment.
  Interventions: Other: Functional Brain Imaging and neurobehavioural tasks

INTERVENTIONS:
Other: Functional Brain Imaging and neurobehavioural tasks — Combination of 3 neurobehavioural tasks:
  Task 1 consists in subjective value rating of 64 food items. Participants are asked to rate how much they would want to eat the presented food item while fMRI (functional magnetic resonance imaging ) scanning is performed.
  Task 2 consists in rating of subjective nutrient factor of the same 64 food items. Participants will answer the following four categorical questions in randomized order for each item: low or high in added sugar/protein/fat and healthy or unhealthy.
  Task 3 consists of a decision-making task. Participants will be presented with two food items (out of the 64 food items), and asked to choose which of the two items they prefer to consume at the end of the experiment.

SUMMARY:
Obesity is currently one of the most substantial health burdens. Due to the production of marked and sustained weight loss, bariatric surgery is an increasingly used therapeutic modality to combat obesity and its comorbidities. Surgical rearrangement of the gastrointestinal tract remarkably alters metabolism and hormones acting on neurological and hypothalamic signalling involved in food decision-making and eating behaviour. In this context, many patients who underwent bariatric surgery self-report changes in appetite, satiety and food preferences. Furthermore, new gut hormone-based (e.g. GLP1-receptor agonist or GLP-1-RA) pharmacotherapies which mimic the effect of bariatric surgery show impressive efficacy on weight reduction by modulation of food behaviour. However, the mechanisms of such functional changes, and how they relate to food decision-making remain unknown.

In this project, the investigators propose a novel approach to unravel the effect of obesity treatments (surgical and non-surgical) on the neural coding of nutritional attributes and its impact on dietary choices using a combination of brain imaging, computational modelling of food behaviour and assessment of eating and food purchase behaviour in daily life.

DETAILED DESCRIPTION:
The overall aim of this project is to elucidate the neurobehavioural underpinnings of food behaviour among obese adults and how food behavior is altered by different obesity treatments.To this end, the study consists of an experimental setting combining neurobehavioural tasks, computational modelling and functional brain imaging.

The main objective of Part 1 of the BrainFood-project is to elucidate if neural coding and food behaviour differ between obese adults and lean adults. The investigators hypothesize that subjective neural processes of nutritional food attributes differ between the obese and control participants, showing an unhealthier pattern among obese participants.

To this aim, the outcomes will be compared between groups (surgery group and control group).

ELIGIBILITY:
Inclusion criteria (all participants):

* Female and male subjects aged 18 years or older
* Proficient German language skills (including written)

Inclusion criteria for Group 1 (pilot protocol):

* Class II-III obesity (BMI≥35kg/m2)
* Planned for bariatric surgery (Roux-en-Y gastric bypass)

Inclusion criteria for Group 1 (refined protocol):

* BMI≥30kg/m2 or BMI≥28kg/m2 with adiposity-related comorbidities (prediabetes, type 2 diabetes mellitus, hypertension, dyslipidemia)
* Referred for obesity treatment (surgical or non-surgical)

Inclusion criteria for Group 2 (pilot and refined protocols):

* Normal body weight (BMI 18.5-24.9kg/m2)
* Absence of evidence of any active or chronic disease as judged by the Clinical Investigator

Exclusion criteria:

* Incapacity to give informed consent
* Previous or current neurological or severe psychiatric illness
* Current or planned pregnancy or breastfeeding
* Claustrophobia
* MRI-contraindications (pacemaker/defibrillator, neurostimulator, drug pump, cochlear implant, heart valve/vascular clips, shunt valve)
* Pilot protocol only: Diabetes according to WHO (World Health Organization ) definition (Fasting plasma glucose ≥7.0mmol/l, random plasma glucose ≥11.1mmol/l, HbA1c ≥6.5%)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Pilot protocol:
  5 obese adults planned for bariatric surgery (Group 1) will be recruited by referral from our outpatient endocrine clinic and collaborating Centres of Excellence for Metabolic Surgery.
  5 lean healthy adults (Group 2) matched for age-, sex- and education will serve as a control group and will be recruited through advertisement according to guidelines from swissethics.
  Refined protocol:
  20 obese adults planned for obesity treatment (Group 1) will be recruited by referral from our outpatient endocrine clinic and collaborating Centres of Excellence for Metabolic Surgery.
  20 lean healthy adults (Group 2) matched for age and sex will serve as a control group and will be recruited through advertisement according to guidelines from swissethics.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2021-04-12 (Actual); Primary Completion 2022-09-05 (Actual); Study Completion 2022-09-05 (Actual)

PRIMARY OUTCOMES:
Representational similarity analysis to assess neural encoding of food attributes | Continuously while participants perform the tasks (during 2.5 hours)
  Representational similarity analysis is used to analyse the correlation between a voxel-wise representational dissimilarity matrix and a behavioural representational dissimilarity matrix. The correlation of the activity of each voxel for each pair of food items is used to define the voxel-wise representational dissimilarity matrix. Similarly, the correlation of the subjective ratings for each pair of food items is used to define the behavioural representational dissimilarity matrix. The correlation between the voxel-wise representational dissimilarity matrix and the behavioural representational dissimilarity matrix is then assessed to determine if the voxels are encoding the food attributes.
Nutrient factor weights | Continuously while participants perform the tasks (during 2.5 hours)
  The nutrient factor weights are estimated using a linear regression with the subjective value ratings as dependent variable and nutrient factors ratings as independent variables and using a logistic regression with the choice as a dependent variable and the nutrient factor ratings as independent variables.

SECONDARY OUTCOMES:
Differences in activity in neural areas involved in self-control and valuation (Dorsolateral prefrontal cortex (dlPFC), ventromedial prefrontal cortex (vmPFC), orbitofrontal cortex (OFC), anterior cingulate cortex (ACC), insula, hippocampus) | Continuously while participants perform the tasks (during 2.5 hours)
  Activity in the neural areas will be compared between groups

CONTACTS AND LOCATIONS:
Overall Officials: Lia Bally, MD, PhD, Principal Investigator — University Hospital Bern & University of Bern
Locations (1):
- Department of Diabetes, Endocrinology, Clinical Nutrition and Metabolism, Inselspital, Bern University Hospital, Bern, Switzerland

IPD SHARING:
Plan to Share IPD: Undecided
To support the development of transparent and open science, the data collected during this study can be published in open science repositories (e.g., Open Science Framework) or with the research articles after acceptance of the research articles. The data will be pseudo-anonymized prior to their publication and the faces will be removed from MRI scans to ensure anonymity.